CLINICAL TRIAL: NCT04674267
Title: Resilience and Equity in Aging, Cancer, and Health (REACH): Promoting Physical Resilience and Cancer Care Equity for Adults Age 70 and Older Diagnosed With Gastrointestinal Malignancy
Brief Title: Resilience and Equity in Aging, Cancer, and Health (REACH)
Acronym: REACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nadine McCleary, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-275
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Gastric Cancer; Colon Cancer; Esophageal Cancer; Rectal Cancer; Pancreatic Cancer; Gastrointestinal Cancer
Keywords: Gastrointestinal cancer
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Rectal Neoplasms; Pancreatic Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Phase - Geriatric Co-Management (Experimental): Eligible older adults age 70 and older who score "Pre-Frail" or "Frail" will be randomized 2:1 to be offered to meet with a study geriatrician for geriatric co-management in addition to their standard oncology care. Study geriatrician will assist with management of symptoms, additional comorbidities, polypharmacy, and social/emotional concerns in addition to physical care. Geriatrician can make referrals and recommendations for additional supportive services that may be beneficial for more vulnerable older adult patients.
  Interventions: Other: Phase 2 Intervention - Geriatric Co-Management
- Intervention Phase - Standard Oncology Care (No Intervention): This arm is for those older adult patients (age 70+) who score as "Pre-Frail" or "Frail" in the fitness assessment questionnaire and are NOT randomized to meet with the study geriatrician. These patients will be followed for the duration of the study as they proceed with their usual oncology care. Study team will evaluate a number of different measures and outcomes, the primary one being unplanned emergency and hospital visits during the course of the study.

INTERVENTIONS:
Other: Phase 2 Intervention - Geriatric Co-Management — Participants will complete an electronic fitness assessment questionnaire - once completed, they will receive a score of "Robust", "Pre-Frail" or "Frail". Those who are "Pre-frail" or "Frail" will be randomized to meet with a study geriatrician for geriatric co-management in addition to usual oncology care. All participants will be followed for a duration of 1 year.
  Arms: Intervention Phase - Geriatric Co-Management

SUMMARY:
The purpose of this multi-phase research study is to understand how consultation of cancer care with a geriatrician can best improve outcomes for older adults with gastrointestinal malignancies.

DETAILED DESCRIPTION:
This research study will be conducted in three phases:

* Phase 1 - Needs assessment and implementation plan
* Phase 2 - Pilot Intervention
* Phase 3 - Expanded Clinical Trial

  * Please note Phase 2 - Pilot Intervention and Phase 3 - Expanded Clinical Trial will be added to the clinicaltrials.gov record once Institutional Review Board (IRB) approved.

Phase 1 is composed of three aims and will inform the subsequent two phases:.

* Aim 1: To evaluate the perceived needs of Older Adults diagnosed with gastrointestinal malignancies, caregivers, staff, and faculty to characterize the implementation setting for a geriatric consultation.
* Aim 2: To refine the proposed REACH program implementation plan based on qualitative feedback provided by Older Adult (OA) patients, their identified caregivers, staff, and faculty.
* Aim 3: Determine the patient, demographic, social determinants, clinical and disease characteristics of Older Adults (OA) associated with ED visits/hospitalization following initial oncology consultation at DF/BWCC in year 2019.
* Phase 2 intervention has started as of January 2022 following IRB approval. Study team has begun recruiting participants into Phase 2 intervention of REACH study starting in January 2022. Participants approached by REACH coordinator for consenting and enrollment after their initial consult visit at Dana-Farber/Brigham and Women's Cancer Center (DF/BWCC). Participants are then asked to complete an electronic fitness assessment (EFA) that is sent to them via Patient Gateway. Participants complete this questionnaire and receive a score of "Robust", "Pre-frail", or "Frail" - those who score "Pre-frail" or "Frail" will be randomized to meet with a study geriatrician for geriatric co-management intervention alongside their standard oncology care. All enrolled participants will be followed for a duration of 1 year as they are continuing care at DF/BWCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are age 70+ at time of initial consult at DF/BWCC
* Diagnosed with a gastrointestinal cancer, including: cancers of the esophagus, stomach, pancreas, liver, bile duct, ampulla, colon, rectum, or anus, as well as neuroendocrine tumors.
* Continuing care at DF/BWCC beyond initial consult visit
* English and Spanish-speaking

Exclusion Criteria:

* Patients less than age 70 at time of initial consultation appointment with DF/BWCC.
* Patients who are not continuing care at DF/BWCC beyond first consult visit.
* Not proficient in English or Spanish
* Patient who are not considered appropriate for enrollment due to complex medical, social, or other situation as determined by their primary oncology team.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 257 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of electronic fitness assessment questionnaire (developed from Comprehensive Geriatric Assessment tool) | 1 year
  EFA questionnaire deployed to older adult patients age 70+ in the REACH study. Feasibility will be determined by the proportion of participants who consent to complete the electronic fitness assessment. The intervention will be considered feasible if 70% of participants consent to complete the fitness assessment.
Acceptability of electronic fitness assessment questionnaire | 1 year
  Acceptability of electronic fitness assessment questionnaire via the Patient Portal or internet-enabled device following second clinic visit among older adults diagnosed with gastrointestinal cancer seeking consultation at DF/BWCC for medical, radiation, or surgical oncology. Acceptability will be determined by the proportion of participants who fully complete the EFA. The intervention will be considered acceptable if 60% of enrolled participants fully complete the EFA within 14 days of enrollment.
Association of geriatric consultation with number of unplanned ED visits/hospitalizations among older adult participants | 1 year
  Association of geriatrician consult with number of ED visits/hospitalizations among older adults diagnosed with gastrointestinal cancer randomized to the geriatric consultation intervention. Randomization will be essential to evaluate the efficacy of geriatric consultation intervention in impacting unplanned ED visits and hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine J McCleary, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu